CLINICAL TRIAL: NCT02117089
Title: Biomechatronic System Using Voluntary Motor Effort (VME)-Driven Neuromuscular Electrical Stimulation (NMES) for Upper Limb Rehabilitation
Brief Title: Upper Limb Rehabilitation After Stroke Assisted With a Hybrid Electrical Stimulation (ES)-Robot System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Xiaoling Hu, Doctor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITS/033/12; ITS/033/12 (Other Grant/Funding Number: Innovation and Technology Commission of Hong Kong)
Record Dates: First submitted 2014-04-10; First posted 2014-04-17 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device-assisted rehabilitation (Experimental)
  Interventions: Device: Electrical Stimulation; Rehabilitation Robot

INTERVENTIONS:
Device: Electrical Stimulation; Rehabilitation Robot — The recruited subjects will receive 20-session device assisted upper limb training with an intensity of 3 to 5 sessions/week, which will be finished within 7 consecutive weeks. In each session, the subjects will conduct the system assisted and task-oriented upper limb training for 1.5 hours.

SUMMARY:
The purpose of this study is to investigate the combined training effectiveness of mechanical robot and neuromuscular electrical stimulation on upper limb rehabilitation after stroke.

ELIGIBILITY:
Inclusion Criteria:

The recruited subjects will

* have unilateral ischemic brain injury or intracerebral hemorrhage at least 6 months after the onset of single stroke
* have moderate level of motor impairment in the affected upper limb, assessed by Fugl-Meyer Assessment (9<shoulder/elbow<27; 6<wrist/hand<18)
* have enough cognition to be able to follow the training protocol as assessed by Mini-metal State Examination (MMSE>21)
* have detectable EMG signals (3 times of the standard deviation above the baseline) from the upper limb muscles.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2013-10; Primary Completion 2024-09 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment Scale after training | 1) up to 7 weeks, 2) 3 months after participants finish the training
  The Fugl-Meyer Assessment Scale for upper limb measures the voluntary motor function on the shoulder, the elbow, the wrist and hand. The full score ranges from 0 to 66. It can be further separated into two subscores, i.e., shoulder/elbow (0-42) and wrist/hand (0-24). The higher the score, the better is the related motor function.
Change in Modified Ashworth Scale after training | 1) up to 7 weeks, 2) 3 months after participants finish the training
  The Modified Ashworth Scale measures the resistance of a joint during passive motion, which indicates the muscle spasticity related to the joint motion, particularly the flexors. The Modified Ashworth Scale has six levels, i.e., 0, 1, 1+, 2, 3, 4. The higher value is related to a higher joint resistance, i.e., higher muscle spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoling Hu, Ph.D., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China

REFERENCES:
- [Derived] Guo Z, Zhou S, Ji K, Zhuang Y, Song J, Nam C, Hu X, Zheng Y. Corticomuscular integrated representation of voluntary motor effort in robotic control for wrist-hand rehabilitation after stroke. J Neural Eng. 2022 Mar 9;19(2). doi: 10.1088/1741-2552/ac5757. PMID 35193124
- [Derived] Ye F, Yang B, Nam C, Xie Y, Chen F, Hu X. A Data-Driven Investigation on Surface Electromyography Based Clinical Assessment in Chronic Stroke. Front Neurorobot. 2021 Jul 15;15:648855. doi: 10.3389/fnbot.2021.648855. eCollection 2021. PMID 34335219
- [Derived] Qian Q, Nam C, Guo Z, Huang Y, Hu X, Ng SC, Zheng Y, Poon W. Distal versus proximal - an investigation on different supportive strategies by robots for upper limb rehabilitation after stroke: a randomized controlled trial. J Neuroeng Rehabil. 2019 Jun 3;16(1):64. doi: 10.1186/s12984-019-0537-5. PMID 31159822
- [Derived] Nam C, Rong W, Li W, Xie Y, Hu X, Zheng Y. The Effects of Upper-Limb Training Assisted with an Electromyography-Driven Neuromuscular Electrical Stimulation Robotic Hand on Chronic Stroke. Front Neurol. 2017 Dec 14;8:679. doi: 10.3389/fneur.2017.00679. eCollection 2017. PMID 29312116
- [Derived] Qian Q, Hu X, Lai Q, Ng SC, Zheng Y, Poon W. Early Stroke Rehabilitation of the Upper Limb Assisted with an Electromyography-Driven Neuromuscular Electrical Stimulation-Robotic Arm. Front Neurol. 2017 Sep 4;8:447. doi: 10.3389/fneur.2017.00447. eCollection 2017. PMID 28928706
- [Derived] Rong W, Li W, Pang M, Hu J, Wei X, Yang B, Wai H, Zheng X, Hu X. A Neuromuscular Electrical Stimulation (NMES) and robot hybrid system for multi-joint coordinated upper limb rehabilitation after stroke. J Neuroeng Rehabil. 2017 Apr 26;14(1):34. doi: 10.1186/s12984-017-0245-y. PMID 28446181